CLINICAL TRIAL: NCT04655196
Title: A Randomized Controlled Trial to Evaluate the Efficacy of Two Internet-based Self-help Interventions for Loneliness.
Brief Title: Evaluation of the Efficacy of Two Internet-based Self-help Interventions for Loneliness.
Acronym: SOLUS-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOLUS-D
Record Dates: First submitted 2020-11-27; First posted 2020-12-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Loneliness
Keywords: internet-based self-help; loneliness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet-based self-help + weekly feedback by a coach (Experimental): Internet-based self-help on the basis of CBT-interventions, mindfulness and self-compassion to address cognitions, emotions and behavior related to loneliness. The self-help program consists of nine text, audio and video-based sessions, various exercises (e.g., breathing meditation, diaries) and tasks. Participants receive weekly feedback by a coach.
  Interventions: Other: SOLUS-D + weekly feedback by a coach
- Internet-based self-help + weekly automated messages (Experimental): Internet-based self-help on the basis of CBT-interventions, mindfulness and self-compassion to address cognitions, emotions and behavior related to loneliness. The self-help program consists of nine text-, audio- and video-based sessions, various exercises (e.g., breathing meditation, diaries) and tasks. Participants receive weekly automated messages in order to increase motivation.
  Interventions: Other: SOLUS-D + weekly automated messages
- Waiting control group (No Intervention)

INTERVENTIONS:
Other: SOLUS-D + weekly feedback by a coach — internet-based self-help
  Arms: Internet-based self-help + weekly feedback by a coach
Other: SOLUS-D + weekly automated messages — internet-based self-help
  Arms: Internet-based self-help + weekly automated messages

SUMMARY:
In this study, people who suffer from loneliness will be randomized to three study conditions. The first and second group get an account to an internet-based self-help intervention. The first group also receives weekly feedback from a coach and the second group receives an automated email on a weekly basis. The third group is a waiting control group. In all three conditions additional care or treatment is allowed. The aim of the study is to investigate the efficacy of an internet-based self-help intervention to reduce feelings of loneliness compared to a waiting list and the effect of support during the intervention. Assessments are at baseline, 5-week, 10-week, 6-months and 12-months post-randomization. Participants in the waiting control group get also access to the intervention and fill out questionnaires at baseline, 5-week and 10-week post-randomization and get also access to the intervention 10 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Sumscore ≥ 18 on the UCLA Loneliness Scale
* Signed Informed Consent
* Contact information provided in case of emergency
* Internet connection and device to use it (Smartphone, Computer, Tablet)
* Fluent in german language

Exclusion Criteria:

* Acute suicidality
* A current diagnose of substance dependence, a current or previous diagnose of psychotic disorder or bipolar disorder
* A current diagnosis of severe depression (PHQ-9 > 14)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Loneliness | 10-week
  Measured with the UCLA Loneliness Scale, 9-Item Version (UCLA-9). Total score ranging from 1-4 (representing the mean score of all 9 items). Lower scores represent less loneliness and a more favourable outcome.

SECONDARY OUTCOMES:
Depressive Symptoms | Baseline, 5-week, 10-week, 6-months, 12-months
  Measured with the Patient Health Questionnaire (PHQ-9). Total score ranging from 0-27 (representing the sum of each of the 9 individual items). Clinical cut-offs for mild, moderate, moderately severe and severe major depressive disorder are considered to be 5, 10, 15, and 20 points.
Satisfaction with Life | Baseline, 5-week, 10-week, 6-months, 12-months
  Measured with the Satisfaction with Life Scale (SWLS). Total score ranging from 1-7 (representing the mean score of all 5 items). Higher scores indicate higher satisfaction with life.
Misanthropy | Baseline, 10-week, 6-months, 12-months
  Measured with the subscale "Misanthropy" of the Embitterment Scale (BVI). Total score ranging from 0-4 (representing the mean score of all 5 items). Higher scores indicate a higher degree in misanthropy.
Self-Stigma in Loneliness | Baseline, 10-week, 6-months, 12-months
  Measured with the Self-Stigma in Loneliness Questionnaire. Total score ranging from 1-5 (representing the mean score of all 6 items). Higher scores indicate higher self-stigma.
Social Interaction Anxiety | Baseline, 10-week, 6-months, 12-months
  Measured with the Social Interaction Anxiety Scale, 6-Item Version (SIAS-6). Total score ranging from 0-5 (representing the mean score of all 6 items) Higher scores indicate higher social interaction anxiety.
Social Phobia | Baseline, 10-week, 6-months, 12-months
  Measured with the Social Phobia Scale, 6-Item Version (SPS-6). Total score ranging from 0-5 (representing the mean score of all 6 items). Higher scores indicate higher social phobia.
Self-Compassion | Baseline, 10-week, 6-months, 12-months
  Measured with the Sussex Oxford Compassion for the Self Scale (SOCS-S). Total score ranging from 1-5 (representing the mean score of all 20 items). Higher scores indicate higher self-compassion.
Social Network | Baseline, 10-week, 6-months, 12-months
  Measured with the Social Network Index (SNI). Network Diversity ranging from 1-8 (representing the number of social roles in which the respondent has regular contact with at least one person). Higher scores indicate a more diverse social network. Number of people in Social Network ranging from 0 to infinity. Higher scores indicate a larger social network.
Diagnostic Interview for Mental Disorders, short-version (Mini-DIPS) | Baseline, 6-months
Interpretation and Judgmental Bias | Baseline, 5-week, 10-week, 6-months, 12-months
  Measured with the Interpretation and Judgmental Questionnaire (IJQ). The interpretation score ranges from 1-4 (representing the chosen likelihood of the profoundly negative alternative). Higher scores indicate more negatively biased processing.
Rejection Sensitivity | Baseline, 5-week, 10-week, 6-months, 12-months
  Measured with the Rejection Sensitivity Questionnaire (A-RSQ). Total score ranging from 1-36 (representing the mean score of the multiplication of the subscales of all 9 items). Higher scores indicate higher rejection sensitivity.
Behavioral-social Avoidance | Baseline, 5-week, 10-week, 6-months, 12-months
  Measured with the "behavioral-social avoidance"-subscale of the Cognitive-Behavioral Avoidance Scale (CBAS). Total score ranging from 1-5 (representing the mean score of all 8 items). Higher scores indicate higher behavioral-social avoidance.
Distress Disclosure | Baseline, 5-week, 10-week, 6-months, 12-months
  Measured with the Distress Disclosure Index (DDI). Total score ranging from 1-5 (representing the mean score of all 12 items). Higher scores indicate higher levels of distress disclosure.
Authenticity | Baseline, 5-week, 10-week, 6-months, 12-months
  Measured with the Kernis-Goldman Authenticity Inventory - Short Form (KGAI-SF). Total score ranging from 1-5 (representing the mean score of all 20 items). Higher scores indicate less authenticity.
Negative Effects | 10-week
  Measured with the Inventory for the Assessment of Negative Effects of Psychotherapy (INEP). Total score ranging from -3-3 (representing the mean score of all items). Higher scores indicate less unfavourable effects of psychotherapy.
Client Satisfaction | 10-week
  Measured with the Client Satisfaction Questionnaire (ZUF-8). Total score ranging from 1-4 (representing the mean score of all 8 items). Higher scores indicate higher client satisfaction.
System Usability | 10-week
  Measured with the System Usability Scale (SUS). Total score ranging from 0-100 (representing the sum score multiplied by 2.5). Higher scores indicate higher perceived usability.
Self-esteem | Baseline, 10-week
  Measured with the Rosenberg Self-Esteem Scale (RSES). Total score ranging from 0-30 (representing the sum of each of the 10 individual items). Higher scores indicate higher self-esteem.
Self-determined motivation for solitude | Baseline, 10-week
  Measured with the subscale "self-determined motivation for solitude" of the Motivation for Solitude Scale - Short Form (MSS-SF). Total score ranging from 1-4 (representing the mean score of all 8 items). Higher scores indicate higher self-determined motivation for solitude.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Krieger, PD Dr., Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Seewer N, Skoko A, Kall A, Andersson G, Luhmann M, Berger T, Krieger T. Efficacy of an Internet-based self-help intervention with human guidance or automated messages to alleviate loneliness: a three-armed randomized controlled trial. Sci Rep. 2024 Mar 19;14(1):6569. doi: 10.1038/s41598-024-57254-0. PMID 38503870
- [Derived] Seewer N, Skoko A, Kall A, Andersson G, Luhmann M, Berger T, Krieger T. Evaluating the Efficacy of a Guided and Unguided Internet-Based Self-help Intervention for Chronic Loneliness: Protocol for a 3-Arm Randomized Controlled Trial. JMIR Res Protoc. 2022 Jul 22;11(7):e36358. doi: 10.2196/36358. PMID 35867403